CLINICAL TRIAL: NCT05357326
Title: Multi-centered Clinical Trial on Myopia Intervention in Children and Adolescents and Establishment of a Precise Intervention Model Based on Deep Learning
Brief Title: Myopia Intervention in Children and Adolescents and Establishment of a Precise Intervention Model
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Eye Disease Prevention and Treatment Center (Other)
Collaborators: Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHYB2021003
Record Dates: First submitted 2021-08-09; First posted 2022-05-02 (Actual); Last update posted 2022-05-02 (Actual); Status verified 2021-08

CONDITIONS: Myopia
Keywords: myopia progression; atropine; orthokeratology
MeSH Terms: conditions — Myopia | interventions — Atropine; Ophthalmic Solutions

STUDY DESIGN:
Intervention Model Description: Children are randomly allocated into three groups: 0.01% atropine, 0.04% atropine and orthokeratology, each group includes 62 children.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 0.01% atropine (Active Comparator): use atropine sulfate 0.01% eye drop every night before sleep for two years
  Interventions: Drug: Atropine Sulfate 0.01% Eye Drop
- 0.04% atropine (Experimental): use atropine sulfate 0.04% eye drop every night before sleep for two years
  Interventions: Drug: Atropine Sulfate 0.04% Eye Drop
- orthokeratology (Experimental): wear orthokeratology lens every night for two years
  Interventions: Device: Orthokeratology

INTERVENTIONS:
Drug: Atropine Sulfate 0.01% Eye Drop — use one drop into subconjunctiva
  Arms: 0.01% atropine
Device: Orthokeratology — wear orthokeratology at night while sleeping
  Arms: orthokeratology
Drug: Atropine Sulfate 0.04% Eye Drop — use one drop into subconjunctiva
  Arms: 0.04% atropine

SUMMARY:
Investigators are going to conduct a multi-centered randomized clinical trial that myopic children are randomly allocated into three groups: 0.01% atropine， 0.04% atropine and orthokeratology in order to evaluate the efficacy and side effects of different intervention methods and establish a risk factor model to predict the efficacy of myopia intervention, and to provide precise intervention plans and clinical decisions for the control of myopia.

DETAILED DESCRIPTION:
Investigators are going to conduct a multi-centered randomized clinical trial that myopic children are randomly allocated into three groups: 0.01% atropine， 0.04% atropine and orthokeratology in order to evaluate the efficacy and side effects of different intervention methods and establish a risk factor model to predict the efficacy of myopia intervention, and to provide precise intervention plans and clinical decisions for the control of myopia.

ELIGIBILITY:
Inclusion Criteria:

* children aged from 8-15 years old;
* children with spherical degree ranged from -1.0D to -4.0D, cylindrical degree less than -1.50D, astigmatism with the rule less than -1.25D, astigmatism with other axial distribution less than -0.50, anisometropia less than -1.50D;
* children with BCVA less than 0.1 LogMAR for both eyes;
* children without other eye diseases except for ametropia

Exclusion Criteria:

* children with other eye diseases: amblyopia, strabismus, eye trauma, etc;
* children with cycloplegia contradictions;
* children who have used atropine or orthokeratology;
* children who are severly allergic with atropine;
* children who are using other eye drops for treatment;
* children who have contraindications to orthokeratology or cannot cooperate with it;
* children with severe heart, lung, liver and kidney diseases

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 186 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2023-07-01 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
spherical equivalent progression in over two years | 2 years
  equals sphere +1/2 cylinder
axial length change over two years | 2 years
  measured by IOL-Master

SECONDARY OUTCOMES:
lens power change over two years | 2 years
  calculated by Bennett-Rabetts formula
choroidal thickness change over two years | 2 years
  measured by SS-OCT
choroidal blood flow density change over two years | 2 years
  measured by OCTA
anterior chamber depth change over two years | 2 years
  measured by IOL-Master
intraocular pressure change over two years | 2 years
  measured by a non-contact tonometer
corneal topography change over two years | 2 years
  measured by Pentacam

CONTACTS AND LOCATIONS:
Overall Officials: Jianfeng Zhu, Study Chair — Shanghai General Hospital, Shanghai Jiao Tong University School of Medicine
Locations (1):
- Jianfeng Zhu, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xu H, Chen M, Ye L, Shu Q, Peng Y, Liang X, Yu T, Ji Y, Li S, Shen Q, He J, Li L, Zhu J, Xu X. Orthokeratology, 0.04% Atropine, and 0.01% Atropine for Myopia Control: A Randomized Clinical Trial. JAMA Ophthalmol. 2025 Jul 24;143(9):731-8. doi: 10.1001/jamaophthalmol.2025.2321. Online ahead of print. PMID 40705323